CLINICAL TRIAL: NCT03571061
Title: Comparisons of Sigmoid-colon Water Immersion, the Whole Colon Water Immersion and Carbon Dioxide (CO2) Insufflation on Cecal Intubation Time in Potentially Difficult Colonoscopy by Difficult Colonoscopy Score(DCS) >1.
Brief Title: Comparisons of SWI, WWI and CI in Potentially Difficult Colonoscopy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: SWI
Record Dates: First submitted 2018-05-28; First posted 2018-06-27 (Actual); Last update posted 2019-01-02 (Actual); Status verified 2018-04

CONDITIONS: Colonoscopy
Keywords: water-aided colonoscopy; difficult colonoscopy
MeSH Terms: interventions — Carbon Dioxide; Insufflation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- whole colon water immersion group (Active Comparator): whole colon water immersion group: the air supply was turn off until the cecum was reached. For adequate lumen distention to advance the colonoscope tip, warm water which stored in 1L bottles and maintained 37°C with a water bath, was instilled intermittently into the colon through the auxiliary working channel of colonoscope using a footswitch-controlled flushing pump
  Interventions: Procedure: whole colon water immersion and sigmoid water immersion
- sigmoid water immersion group (Experimental): sigmoid water immersion group: air pump would be turned off and the procedure would be switched from water immersion method to air insufflation method after successful passage through the descending sigmoid junction.
  Interventions: Procedure: whole colon water immersion and sigmoid water immersion
- carbon dioxide (CO2) insufflation (Placebo Comparator): carbon dioxide (CO2) insufflation group: carbon dioxide (CO2) was insufflated through out the whole procedure for advancement and inspection when needed.
  Interventions: Procedure: whole colon water immersion and sigmoid water immersion

INTERVENTIONS:
Procedure: whole colon water immersion and sigmoid water immersion — we chose water immersion method instead of the triaditional method of carbon dioxide (CO2) insufflation.
  Other Names: carbon dioxide (CO2) insufflation

SUMMARY:
Colonoscopy insertion is technically challenging, time-consuming, and painful, especially for the sigmoid. It is reported that the difficult colonoscopy score (DCS) >1 can predict the difficulty during colonoscopy. Patients with DCS>1 had longer insertion time, higher pain score and needed more abdominal compression and position changes. As reported, water-aided method colonoscopy examination is an important and useful method because it reduces discomfort and increases cecal intubation rate compared with usual air insufflation method. But a longer time was consumed for scope insertion and cecal intubation in the traditional water-aided method colonscopy(the whole water immersion). To avoid these disadvantages ,we modified whole colon water immersion(WWI) method to the sigmoid colon water immersion(SWI), where the most difficult and painful part of colonoscopy resides. If water immersion is limited to the sigmoid colon in such patients, would it be more efficient and less time consuming?

The aim of this study was to investigate the application of water-aided method on cecal intubation time in potentially difficult colonoscopy. This prospective, randomized controlled study allocated patients who's difficult colonoscopy score(DCS) >1 (18-80 years) to sigmoid-colon water immersion(SWI), whole colon water immersion(WWI) or carbon dioxide (CO2) insufflation (CI) group (1:1:1). The primary outcome was cecal intubation time. The secondary outcomes included the maximum pain score (0=none,10=most severe) during the insertion phase in left, transverse and right colon; cecal intubation rate; adenoma detection rate(ADR); bowel preparation quality; withdrawal time(from cecum to rectum excluding time for biopsy and polypectomy); willingness to undergo a repeat unsedated colonoscopy; number of abdominal compressions, position change during the insertion. Patients were educated to understand the meaning of visual analogue scale (VAS) (0 = no pain, 10 = most severe) and to report their maximum pain scores during the insertion through each colonic segment. Descriptive statistics were used to summarize demographic and baseline data. Analyses were performed with SPSS software version 24.0 for Windows (SPSS Inc, IBM Company).

DETAILED DESCRIPTION:
Introduction: Colonoscopy insertion is technically challenging, time-consuming, and painful, especially for the sigmoid. Many factors have been found to affect the difficulty of colonoscope insertion, such as age, gender, body mass index, history of abdominal surgery and operator ect. It is reported that the difficult colonoscopy score (DCS) >1 can predict the difficulty during colonoscopy. DCS=1*A(1 if age≥65y, 0 if <65y) + 2*B (1 if BMI <18.5, 0 if BMI≥18.5) + 1*C (1 if colonoscopist is junior, 0 if senior)+ 1*S(1 if sleep quality was fair or bad, 0 if excellent or good). Patients with DCS>1 had longer insertion time, higher pain score and needed more abdominal compression and position changes. For these potentially difficult cases we can use special intubation techniques such as water-aided or cap-assisted method at the very start to avoid of excessive insertion time, increased discomfort and even unnecessary adverse events.

Water-aided method colonoscopy examination is an important and useful method because it reduces discomfort and increases cecal intubation rate compared with usual air insufflation method. This examination is usually performed using two different methods: water immersion and water exchange. In the water immersion method, the water is infused into the colon beginning with the scope inserted into the anus during examination until the scope reaches the cecum. The water is evacuated during colonoscope withdrawal. In the water exchange method, the water is evacuated during colonoscope advancement until the cecum is reached. The air pump of the endoscopy machine is turned off during examination in both procedures. The aim of this study was to investigate the application of water-aided method on cecal intubation time in potentially difficult colonoscopy. We chose water immersion method rather than water exchange for this evaluation because water immersion, characterized by suction removal of the infused water predominantly during withdrawal, is more appropriate for reducing the cecal intubation time. Further more ,as reported, left-colon water exchange(LWE) shorten the insertion time while preserving the benefits of whole colon water exchange(WWE). We modified whole colon water immersion(WWI) method to the sigmoid colon water immersion(SWI), where the most difficult and painful part of colonoscopy resides. If water immersion is limited to the sigmoid colon in such patients, would it be more efficient and less time consuming? Methods:This prospective, randomized controlled study allocated patients who's difficult colonoscopy score(DCS) >1 (18-80 years) to sigmoid-colon water immersion(SWI), whole colon water immersion(WWI) or carbon dioxide (CO2) insufflation (CI) group (1:1:1). Patients were randomized to SWI, WWI or CI group according to a computer-generated randomization list in 1:1:1 ratio. Group assignments were revealed immediately before the insertion of colonoscopy by a researcher , who did not participate in data collection and data analysis. The monitor screen was placed over the head of patients to keep them from knowing the insertion method. Endoscopists and assisting nurses were not blinded. For the bowel preparation, all patients were instructed to take low-fiber diet for lunch and clear liquid diets for dinner the day before examination. They ingested 2L of PEG powder (WanHe Pharmaceutical Co, Shenzhen, China) diluted with water within 2 h, between 4:00 AM and 5:00 AM on the day of the examination. Those with chronic constipation received an additional 2L of PEG solution on the evening prior to the examination. Drinking more clear water and pacing back and forth after purgatives were encouraged to enhance laxative effect. The time interval between preparation and colonoscopy was limited to less than 5 h to ensure the quality of bowel preparation.

Endoscopic procedure Two endoscopists (WBH and YJ) with extensive experience in both air (>5000) and water methods (>500) performed the colonoscopies. The standard adult colonoscope (EC-600WM, Fujinon, Beijing) was used. Patients were placed in the left lateral position at the beginning of the procedure. Maneuvers such as abdominal compression and position change were implemented if needed (e.g. when looping, paradoxical movement or lack of advancement occurred). Successful cecal intubation was confirmed by the visualization of appendiceal orifice or ileocecal valve with the tip of the colonoscope touching the base of the cecum. For the AI method, air was insufflated through out the whole procedure for advancement and inspection when needed. In the WWI method,the air supply was turn off until the cecum was reached. For adequate lumen distention to advance the colonoscope tip, warm water which stored in 1L bottles and maintained 37°C with a water bath, was instilled intermittently into the colon through the auxiliary working channel of colonoscope using a footswitch-controlled flushing pump. For patients allocated to SWI group, air pump would be turned off and the procedure would be switched from water immersion method to air insufflation method after successful passage through the descending sigmoid junction.

The primary outcome was cecal intubation time. The secondary outcomes included the maximum pain score (0=none,10=most severe) during the insertion phase in left, transverse and right colon; cecal intubation rate; adenoma detection rate (ADR); bowel preparation quality; withdrawal time(from cecum to rectum excluding time for biopsy and polypectomy); willingness to undergo a repeat unsedated colonoscopy; number of abdominal compressions, position change during the insert.

Descriptive statistics were used to summarize demographic and baseline data. Quantitative variables are expressed as means and standard deviations and analyzed by ANOVA followed by Bonferroni test for multiple comparisons. Categorical variables in three groups were compared with chi-square test or Fisher exact test when appropriate. All p-Values were two-sided and those < 0.05 were considered to be significant. Analyses were performed with SPSS software version 24.0 for Windows (SPSS Inc, IBM Company).

ELIGIBILITY:
Inclusion Criteria:

1. patients undergoing diagnostic, screening or surveillance colonoscopy
2. their difficult colonoscopy score(DCS) >1. DCS=1*A(1 if age≥65y, 0 if <65y) + 2*B (1 if BMI <18.5, 0 if BMI≥18.5) + 1*C(1 if colonoscopist is junior, 0 if senior)+ 1*S(1 if sleep quality was fair or bad, 0 if excellent or good).

Exclusion Criteria:

1. history of colorectal resection;
2. sedated colonoscopy;
3. severe colonic stricture or obstructing tumor known before colonoscopy;
4. current pregnancy;
5. hemodynamic instability
6. inability to provide informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2018-11-26 (Actual); Study Completion 2018-12-26 (Actual)

PRIMARY OUTCOMES:
cecal intubation time | 3 months
  the time the colonoscope advanced from the anus to the cecum

SECONDARY OUTCOMES:
maximum pain score | 3 months
  0=none, 10=most severe
withdrawal time | 3 months
  from cecum to rectum excluding time for biopy and polypectomy

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen People's Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jia H, Wang L, Luo H, Yao S, Wang X, Zhang L, Huang R, Liu Z, Kang X, Pan Y, Guo X. Difficult colonoscopy score identifies the difficult patients undergoing unsedated colonoscopy. BMC Gastroenterol. 2015 Apr 9;15:46. doi: 10.1186/s12876-015-0273-7. PMID 25886845
- [Background] Zhang Z, Wu Y, Sun G, Zhang J, Li J, Qiu C, Zheng X, Wang B, Yang L, Wang X. Bayesian network meta-analysis: Efficacy of air insufflation, CO2 insufflation, water exchange, and water immersion in colonoscopy. Dig Endosc. 2018 May;30(3):321-331. doi: 10.1111/den.13012. Epub 2018 Feb 5. PMID 29334136
- [Background] Cadoni S, Leung FW. Water-Assisted Colonoscopy. Curr Treat Options Gastroenterol. 2017 Mar;15(1):135-154. doi: 10.1007/s11938-017-0119-1. PMID 28205108
- [Background] Wang X, Luo H, Xiang Y, Leung FW, Wang L, Zhang L, Liu Z, Wu K, Fan D, Pan Y, Guo X. Left-colon water exchange preserves the benefits of whole colon water exchange at reduced cecal intubation time conferring significant advantage in diagnostic colonoscopy - a prospective, randomized controlled trial. Scand J Gastroenterol. 2015 Jul;50(7):916-23. doi: 10.3109/00365521.2015.1010569. Epub 2015 Feb 1. PMID 25639787
- [Background] von Renteln D, Robertson DJ, Bensen S, Pohl H. Prolonged cecal insertion time is associated with decreased adenoma detection. Gastrointest Endosc. 2017 Mar;85(3):574-580. doi: 10.1016/j.gie.2016.08.021. Epub 2016 Aug 31. PMID 27590962